CLINICAL TRIAL: NCT00998036
Title: Phase I Study of Combined Temsirolimus, Erlotinib and Cisplatin in Advanced Solid Tumors
Brief Title: Study of Temsirolimus, Erlotinib and Cisplatin in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Kevin Kalinsky, Assistant Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD8279
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Triple Negative Breast Cancer
Keywords: TNBC; Temsirolimus; Erlotinib; Cisplatin; Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — temsirolimus; Cisplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Temsirolimus, cisplatin, erlotinib (Experimental): Cisplatin and temsirolimus will be administered weekly on days one and eight of a three week cycle. Erlotinib will be taken by mouth daily.
  Interventions: Drug: Temsirolimus; Drug: Cisplatin; Drug: Erlotinib

INTERVENTIONS:
Drug: Temsirolimus — Temsirolimus will be administered intravenously weekly on days one and eight of a three week cycle. Temsirolimus will not be given on week three (usually dosed weekly) for increased tolerability given its possible plasma accumulation during week three. Temsirolimus will be given second over a 30 minute infusion during posthydration.
  Dose escalation will follow the standard 3 by 3 design with three set dosing levels.
  Dose Level 1: Temsirolimus 15mg
  Dose Level 2: Temsirolimus 15mg
  Dose Level 3: Temsirolimus 25mg
  Other Names: Torisel
Drug: Cisplatin — Cisplatin at 30mg/m2 will be administered intravenously weekly on days one and eight of a three week cycle. Cisplatin will be given first over a 30 minute infusion with prehydration.
  Other Names: Platinol
Drug: Erlotinib — Erlotinib will be taken by mouth daily starting at 100mg. On days of cisplatin and temsirolimus infusions, erlotinib should be taken at least two hours after the beginning of the temsirolimus infusion.
  Dose escalation will follow the standard 3 by 3 design with three set dosing levels.
  Dose Level 1: Erlotinib 100mg
  Dose Level 2: Erlotinib 150mg
  Dose Level 3: Erlotinib 150mg
  Other Names: Tarceva

SUMMARY:
This is a Phase I research study designed to determine the maximum tolerated dose (MTD) of cisplatin, temsirolimus, and erlotinib in combination for treatment in triple negative breast cancer (TNBC) patients.

DETAILED DESCRIPTION:
The stratification of breast cancer patients for treatment targeting either the estrogen receptor (ER) or human epidermal growth factor receptor 2 (HER2) receptor based upon the measurement of ER/progesterone receptor (PR) and HER2 in tumor tissue has changed the treatment of breast cancer. However, the success of this stratification has resulted in the recognition that no effective rational treatment exists for patients that lack these receptors. The term "triple negative breast cancer" (TNBC) has been used to define a class of unresponsive patients, which is based upon their lack of the hormone receptors for estrogen and progesterone and the HER2 oncogene. TNBC represents a form of breast cancer for which no targeted therapy is known.

Thus, identifying and understanding the signaling pathways and receptors that contribute to triple negative tumor growth is of high priority in order to develop therapies analogous to the ones that have already been developed for HER2 and ER.

Available data from Phase I trials have demonstrated that mTOR inhibitors and EGFR inhibitors have been safely given together at doses shown to inhibit their respective targets and Phase II studies are ongoing in advanced renal cell, pancreatic, glioma, and breast (not specifically TNBC) cancers.

The rationale for adding cisplatin to erlotinib and an mTOR inhibitor are many. Cisplatin is a known active cytotoxic against breast cancer. It has non overlapping toxicity with erlotinib and TORC1 mTOR inhibitors and patients are unlikely to have been previously treated with cisplatin. Therefore, as a cytotoxic DNA damaging agent, cisplatin could trigger cell death in a cell whose survival pathways are effectively inhibited by mTOR inhibition and erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic diagnosis of a solid tumor that is not curable with available therapies for which the combination of cisplatin, temsirolimus, and erlotinib is a reasonable treatment.
* Patients with measurable or non-measurable disease are eligible for entry to this study. Tumor markers may be considered non-measurable disease.
* Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. No chemotherapy or radiotherapy may be given within 3 weeks prior to the start of protocol treatment.
* Patients must be ≥18 years old.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0-1
* Life expectancy of greater than 12 weeks.
* Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Required Laboratory Values: absolute neutrophil count (ANC) ≥1,500/mm3, platelets ≥100,000/mm3, hemoglobin ≥9.0 g/dL, total bilirubin ≤1.5 x upper limit of normal (ULN), aspartate transaminase (AST)/alanine transaminase (ALT) ≤3.0 x ULN, alkaline phosphatase ≤2.5 x ULN, creatinine ≤2.0 x ULN OR Patients must have either a normal serum creatinine (<= IULN) OR estimated creatinine clearance 60 ml/min (Cockcroft-Gault formula) within 28 days prior to registration. Prothrombin time (PT)/INR ≤1.5, unless the patient is on full dose warfarin or stable dose of low-molecular-weight (LMW) heparin with a therapeutic INR of >1.5 - ≤3. Patients with triglyceride levels >400 mg/dL can be started on lipid lowering agents and reevaluated within 1 week. If levels go to ≤400 mg/dL, they can be considered for the trial and continue the lipid lowering agents.
* Concomitant Medications: Temsirolimus and Erlotinib are primarily metabolized by CYP3A4. Patients CANNOT be receiving enzyme-inducing or enzyme inhibiting agents listed here: Inhibitors: Amiodarone, Amprenavir, Atazanavir, Chloramphenicol, Clarithromycin, Conivaptan, Cyclosporine, Darunavir, Dasatinib, Delavirdine, Diltiazem, Erythromycin, Fluconazole, Fluoxetine, Fluvoxamine, Fosamprenavir, Imatinib, Indinavir, Isoniazid, Itraconazole, Ketoconazole, Lapatinib, Miconazole, Nefazodone, Nelfinavir, Posaconazole, Ritonavir, Quinupristin, Saquinavir, Tamoxifen, Telithromycin, Troleandomycin, Verapamil, Voriconazole. Inducers: Aminoglutethimide, Bexarotene, Bosentan, Carbamazepine, Efavirenz, Fosphenytoin, Griseofulvin, Modafinil, Nafcillin, Nevirapine, Oxcarbazepine, Phenobarbital, Phenytoin, Primidone, Rifabutin, Rifampin, Rifapentine, St. John's wort, Sulfadimidine, Sulfinpyrazone, Troglitazone, Troleandomycin. All concomitant medications must be recorded. Patients also must agree to refrain from drinking grapefruit juice while on study.
* Sexually Active Patients: For all sexually active patients, the use of adequate contraception (hormonal or barrier method of birth control) will be required prior to study entry and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential.
* Patients must have signed an approved informed consent.

Exclusion Criteria:

* More than 3 prior chemotherapy treatments for metastatic disease.
* Patients receiving anti-retroviral therapy (HAART) for HIV infection because of possible pharmacokinetic interactions.
* Active central nervous system (CNS) disease
* Any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.
* Patients pregnant or nursing.
* Patients who have used tobacco or nicotine products containing medications within the last three months given their significant effect on erlotinib drug levels.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Cisplatin | 6 months
  MTD of the drug as part of combination therapy will be determined.
MTD of Temsirolimus | 6 months
  MTD of the drug as part of combination therapy will be determined.
MTD of Erlotinib | 6 months
  MTD of the drug as part of combination therapy will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kalinksy, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States